CLINICAL TRIAL: NCT05585177
Title: A Randomized Controlled Trial of Growth Hormone to Improve the Clinical Outcome of Assisted Fertility in Young Patients With Decreased Ovarian Reserve
Brief Title: Growth Hormone to Improve the Clinical Outcome of Assisted Fertility in Young Patients With Decreased Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Principal Investigator of Reproductive Medicine Center of The Affiliated Drum Tower Hospital of Nanjing University Medical Scho, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-2022-GH
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormone pretreatment+IVF/ICSI (Experimental): After 3 months of Growth hormone treatment (2 units daily), IVF/ICSI was performed
  Interventions: Drug: Growth hormone
- IVF/ICSI (No Intervention): IVF/ICSI was performed

INTERVENTIONS:
Drug: Growth hormone — 3 months of growth hormone treatment (2 units daily)
  Other Names: IVF/ICSI
  Arms: Growth hormone pretreatment+IVF/ICSI

SUMMARY:
This study was a prospective randomized controlled trial. Patients aged <35 years with decreased clinical reserve function (AFC<5, Follicle stimulating hormone > 10miu/ml, Anti-mullerian hormone < 1.1μg/L) and receiving IVF/ICSI assisted ovulation induction in our hospital were included in this study. After randomization using Excel(Microsoft Corporation, Albuquerque, USA), these patients were divided into two groups. Group A was the experimental group, which was treated with growth hormone for 3 months (2 units per day) before IVF/ICSI. Group B was the control group, which was directly assisted by IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 35 years;
2. AFC≤5
3. Follicle stimulating hormone > 10miu/ml;
4. Anti-mullerian hormone < 1.1μg/L

(2 out of 2-4 items can be met)

Exclusion Criteria:

1. Severe male factors: spermatozoa collected by testicular sperm aspiration (TESA) or percutaneous epididymal sperm aspiration (PESA) was used for intracytoplasmic sperm injection (ICSI) cycle of single spermatozoa;
2. Patients with severe adenomyosis, endometriosis, intrauterine adhesions and other diseases that significantly affect embryo implantation;
3. Diabetes mellitus, insulin resistance;
4. chromosomal karyotype abnormality in either spouse;
5. Any pregnancy or contraindications of assisted reproductive technology;

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of embryos | 4 months
  When at least one dominant follicle reached a diameter of 18 mm or higher, 0.2 mg triptorelin was combined with 10000IU human chorionic gonadotropin as the trigger, and ovarian puncture was performed 36 hours later for oocyte retrieval. The number of embryos formed after three days of combined sperm and egg culture in vitro was recorded.

SECONDARY OUTCOMES:
The number of oocytes retrieved | 4 months
  When at least one dominant follicle reached a diameter of 18 mm or higher, 0.2 mg triptorelin was combined with 10000IU human chorionic gonadotropin as the trigger, and ovarian puncture was performed 36 hours later for oocyte retrieval. The number of oocytes retrieved was recorded.
Clinical pregnancy rate | 5-8months
  Clinical pregnancy was defined as diagnosed by increasing serum concentration of beta-Human chorionic gonadotropin 14 days after embryo transfer, and the subsequent demonstration of an intrauterine gestational sac by ultrasonography on 30 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, PHD, Study Director — The affiliated Drum Towel Hospital of Nanjing University Medical School
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China